CLINICAL TRIAL: NCT06671665
Title: Effect of Manual Therapy on Low Back Pain in Osteopenic Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanan Karamallah Mohamed Abdelkawy, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005212
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Low Back Pain; Osteopenia
MeSH Terms: conditions — Low Back Pain; Bone Diseases, Metabolic | interventions — Calcium Citrate; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium supplementation (Active Comparator): It will consist of 20 postmenopausal women. They will receive calcium supplementation daily for 12 weeks.
  Interventions: Drug: calcium supplementation
- calcium supplementation + manual therapy (Experimental): It will consist of 20 postmenopausal women. They will receive the same calcium supplementation daily in addition to manual therapy (in form of craniosacral technique & general visceral mobilization) for 12 weeks.
  Interventions: Drug: calcium supplementation; Other: Manual therapy

INTERVENTIONS:
Drug: calcium supplementation — Patients in both groups received calcium supplementation in the form of tablets that contain 665 mg calcium citrate. Citrate is easily assimilated and metabolized which provides the maximum benefit of the formula. Dosage: one tablet daily.
  Other Names: 665 mg calcium citrate
Other: Manual therapy — Manual therapy treatment will be in the form of craniosacral techniques and visceral manipulation techniques for 8 sessions in 12 weeks. Sessions will be divided into one session per week for the first 4 weeks then one session every two week for the next 8 weeks. Each session lasts for 45 minutes.
  Arms: calcium supplementation + manual therapy

SUMMARY:
The purpose of this study is to determine the effect of manual therapy on low back pain in osteopenic postmenopausal women.

DETAILED DESCRIPTION:
Women spend nearly one-third of their life in menopause. In this period, besides other comorbid conditions, women suffer from various musculoskeletal disorders also. One such problem is chronic low back pain which is more prevalent in post-menopausal women. This condition affects daily living activities of a person ranging from standing up, walking, bending over, lifting, traveling, social interaction, dressing to sleeping, living with ongoing pain causes depression, anxiety, deterioration in quality of life for women themselves. Despite this, little attention has been paid to pain in the spine/low back ache which are equally prevalent in this period of life.

Although this poses a great medical and socioeconomic challenge to such extent that some researchers call it a lifestyle disease. It is the main cause of absence in the workplace and the 2nd cause of visiting primary health-care professionals. Spine pain has negative psychological consequences as it impairs daily functioning. Therefore, finding an effective method for treatment is important.

Manual treatments are one of the most applied methods within physiotherapy approaches in recent years. Manual treatment (in the form of craniosacral and visceral manipulation) claiming to release the tension of the muscles, ligaments, and fascia in the sacral area and activate central pain inhibitory centers. For this reason, we are conducting the present study with a new view to identify the effects of manual therapy practices in the form of craniosacral and visceral manipulation on pain, function, and BMD of the lumbar region, as well as quality of life in osteopenic post-menopausal women suffering from low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory, sedentary, non-smoking women having natural menopause at least 1 year before participation in the study.
2. Their ages will range from 50 to 60 years old.
3. Their BMI will be > 30 kg/m2.
4. Pain before costal margin and above inferior gluteal fold.
5. Osteopenia.

Exclusion Criteria:

1. Osteoporosis.
2. Having osteoporotic fractures.
3. Having a lumbar surgery previously.
4. Neurological disorder.
5. Known diseases affecting bone quality (hyperthyroidism, hyperparathyroidism, hypercortisolism, etc).
6. Receiving any medical or hormonal therapies that could affect the bone metabolism.
7. Receiving previous manual treatment.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-05-07 (Estimated); Study Completion 2025-06-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of Low back pain severity | 12 weeks
  Pain will be assessed by Visual analog scale (VAS). It is a scale that allows continuous data analysis and uses a 10cm line with 0 (0 = no pain) written at one end and 10 (10 = worst pain) on the other end. Subjects will be asked to place a mark along the line to denote their level of pain.
Measurement of lumbar curvature angle. | 12 weeks
  It will be measured, before and after treatment program, using a flexible ruler. The flexible ruler will be molded to the midline contour of the lumber spine from the spinous process of T12 to S2 to measure the degree of lordosis which carefully traced onto paper using pencil. Then, the lumbar curvature angle will be measured by the equation (theta angle = 4Arctang 2H/L). In this equation, the theta angle represents the magnitude of the lordotic curve, L is a straight line from the first vertebrae to the last vertebrae and the H letter is the distance between the deep point of L line and the lumbar curve.
Assessment of Lumbar Flexion | 12 weeks
  The examiner will stand behind the standing patient to identify the posterior superior iliac spines with thumbs, and then an ink mark will be drawn along the midline of the lumbar spine horizontal to the posterior superior iliac spines. Another ink mark will be made 15 cm above the original mark. The tape measure will be lined up between skin markings. With the tape pressed firmly against the subject's skin and while holding it with fingertips, the distance between superior and inferior skin marks will be measured. Then, the examiner will instruct the patient to bend forward into full lumbar flexion and the new distance between superior and inferior skin marks will be measured. The change in the difference between marks will be used to indicate the amount of lumbar flexion.
Assessment of Lumbar Extension | 12 weeks
  The examiner will follow the same procedure done previously in lumbar flexion except with the instruction. As the examiner will instruct the patient to bend backward into full extension and the new distance between superior and inferior skin marks will be measured as a straight line. The change in the difference between marks will be used to indicate the amount of lumbar extension.
Assessment of Lumbar Lateral bending to the right side | 12 weeks
  Measuring the distance between the tip of the middle finger and the floor when the patient stands upright, heels, buttocks and shoulders against the wall, and bends sideways without lifting the opposite foot off the ground.
Assessment of Lumbar Lateral bending to the left side | 12 weeks
  Measuring the distance between the tip of the middle finger and the floor when the patient stands upright, heels, buttocks and shoulders against the wall, and bends sideways without lifting the opposite foot off the ground.
Assessment of functional disability related to low back pain | 12 weeks
  Functional disability of each patient will be measured using Oswestry disability questionnaire. It is a valid and reliable tool consists of 10 multiple choice questions for back pain; subjects selected one sentence out of six that best describe her pain, higher scores indicated great pain. Scores of minimal disability:(0-20%), Scores of moderate disability: (20%- 40%), Scores of severe disability: (40% - 60%), Scores of crippled subjects: (60% - 80%), and Scores of patients confined to bed (80%-100%).

SECONDARY OUTCOMES:
Measurement of lumbar Bone Mineral Density (BMD) | 12 weeks
  The lumbar BMD of each postmenopausal woman in both groups will be measured before entry into the study to confirm her diagnosis of osteopenia (from -1.1 to -2.49 SD) and also after 12 weeks of treatment, using DEXA, which represents the most preferable method for BMD calculation.
Assessment of quality of life | 12 weeks
  It will be assessed through Short Form 36 Health Survey Questionnaire (SF-36) for both groups before and after the treatment. It comprises eight domain scores including 'physical functioning'. This domain asks respondents to report limitations on ten mobility activities, such as walking specified distances, carrying groceries and bathing or dressing. It is an established and widely used health-related quality of life measure.It consists of ten multiple choice questions for back pain; patient will select one sentence out of six that best describe her pain, higher scores will indicate greater pain and disability. It will be used to measure the level of functional disability due to low back pain. The scores were scaled to a range where 0 denotes the lowest health status and 100 denotes the highest.

CONTACTS AND LOCATIONS:
Overall Officials: Amel M. Yousef, PhD, Study Chair — Professor, Cairo University
Locations (1):
- Cairo University, Giza, Egypt